CLINICAL TRIAL: NCT01923740
Title: A Clinical Evaluation of Absorb™ BVS, the Bioresorbable Vascular Scaffold, in the Treatment of Subjects With de Novo Native Coronary Artery Lesions in Chinese Population
Brief Title: A Clinical Evaluation of Absorb™ Bioresorbable Vascular Scaffold (Absorb™ BVS) System in Chinese Population ~ ABSORB CHINA Randomized Controlled Trial (RCT)
Acronym: ABSORB CHINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-397
Record Dates: First submitted 2013-07-25; First posted 2013-08-16 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Disease; Coronary Stenosis
Keywords: Absorb™ BVS; Angioplasty; Bioabsorbable; BVS; Bioresorbable; Coronary Artery Disease; Coronary Artery Endothelial Responsiveness; Coronary artery restenosis; Coronary artery stenosis; Coronary scaffold; Coronary Stent; Drug eluting stents; Everolimus; Myocardial ischemia; Stent thrombosis; Stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Disease; Coronary Restenosis; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorb BVS System (Experimental): Absorb BVS System: Subjects receiving Absorb BVS System
  Interventions: Device: Absorb BVS System
- XIENCE V EECSS (Active Comparator): XIENCE V EECSS: Subjects receiving XIENCE V
  Interventions: Device: XIENCE V EECSS

INTERVENTIONS:
Device: XIENCE V EECSS — Subjects receiving XIENCE V
  Arms: XIENCE V EECSS
Device: Absorb BVS System — Subjects receiving Absorb BVS System
  Arms: Absorb BVS System

SUMMARY:
To evaluate the safety and efficacy of the Absorb BVS System compared to the XIENCE V Everolimus Eluting Coronary Stent System (EECSS) in the treatment of subjects with ischemic heart disease caused by up to two de novo native coronary artery lesions in separate epicardial vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age at the time of signing the informed consent form.
2. Subject or a legally authorized representative must provide written Informed Consent prior to any study related procedure.
3. Subject must have evidence of myocardial ischemia (e.g., stable angina, unstable angina, post-infarct angina or silent ischemia) suitable for elective percutaneous coronary intervention (PCI). Subjects with stable angina or silent ischemia and < 70% diameter stenosis must have objective sign of ischemia as determined by one of the following, echocardiogram, nuclear scan, ambulatory ECG or stress ECG. In the absence of noninvasive ischemia, fractional flow reserve (FFR) must be done and indicative of ischemia.
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Female subject of childbearing potential does not plan pregnancy for up to 1 year following the index procedure. For a female subject of childbearing potential, a pregnancy test must be performed with negative results known within 14 days (≤14 days) prior to the index procedure per site standard test.
6. Female subject is not breast-feeding at the time of the screening visit and will not be breast-feeding for up to 1 year following the index procedure.
7. Subject agrees to not participate in any other investigational clinical studies for a period of 1 year following the index procedure.

Exclusion Criteria:

1. Any surgery requiring general anesthesia or discontinuation of aspirin and/or P2Y12 inhibitor is planned within 12 months after the index procedure.
2. Subject has a known hypersensitivity or contraindication to device material (cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers) and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid). Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
3. Subject has a known allergic reaction, hypersensitivity or contraindication to:

   1. Aspirin; or
   2. All P2Y12 inhibitors (including clopidogrel and ticlopidine, and prasugrel and ticagrelor when they become available); or
   3. Heparin and bivalirudin.
4. Subject had an acute myocardial infarction (AMI) within 7 days of the index procedure and both creatine kinase (CK) and creatine kinase myocardial-band isoenzyme (CK-MB) have not returned to within normal limits at the time of index procedure.
5. Subject is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
6. Subject has a cardiac arrhythmia as identified at the time of screening which at least one of the following criteria is met:

   1. Subject requires coumadin or any other agent for chronic oral anticoagulation.
   2. Subject likely to become hemodynamically unstable due to their arrhythmia.
   3. Subject has poor survival prognosis due to their arrhythmia.
7. Subject has a known left ventricular ejection fraction (LVEF) < 30% assessed by any quantitative method. LVEF may be obtained within 6 months prior to the procedure for subjects with stable coronary artery disease (CAD). For subjects presenting with acute coronary syndrome (ACS), LVEF must be assessed during the index hospitalization (which may include during the index procedure by contrast left ventriculography) but prior to randomization in order to confirm the subject's eligibility.
8. Subject has received CABG at any time in the past.
9. Subject has undergone prior PCI within the target vessel during the last 12 months or undergone prior PCI within the non-target vessel within 30 days before the index procedure.
10. Subject requires future staged PCI either in target or non-target vessels.
11. Subject has received any solid organ transplants or is on a waiting list for any solid organ transplants.
12. At the time of screening, the subject has a malignancy that is not in remission.
13. Subject is receiving immunosuppressant therapy or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
14. Subject has previously received or is scheduled to receive radiotherapy to coronary artery (vascular brachytherapy), or chest/mediastinum.
15. Subject is receiving or will receive chronic anticoagulation therapy (e.g., coumadin or any other anticoagulation agents).
16. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
17. Subject has a known or documented hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
18. Subject has known renal insufficiency as defined as an estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2 or dialysis at the time of screening.
19. Subject is high risk of bleeding; has a history of bleeding diathesis or coagulopathy; has had a significant gastro-intestinal or significant urinary bleed within the past six months; will refuse blood transfusions.
20. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months or any prior intracranial bleed, any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc.).
21. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion. Note: femoral arterial disease does not exclude the subject if radial or brachial access can be used.
22. Subject has life expectancy < 2 years for any non-cardiac cause or cardiac cause.
23. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
24. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint or protocol-required medications or invasive procedures.

Angiographic Inclusion Criteria

Assessment of angiographic eligibility is per visual assessment by an investigator both for qualitative and quantitative variables. On-line QCA is recommended to be used for appropriately sizing of the vessel. If on-line QCA cannot be used, visual estimation is required.

1. One or two de novo target lesions:

   1. If there is one target lesion, a second non-target lesion may be treated but the non-target lesion must be present in a different epicardial vessel, and must be treated first with a successful, uncomplicated result prior to randomization of the target lesion.
   2. If two target lesions are present, they must be present in different epicardial vessels and both satisfy the angiographic eligibility criteria.
   3. The definition of epicardial vessels means the left anterior descending artery (LAD), the left circumflex artery (LCX), and the right coronary artery (RCA) and their branches. Thus, for example, the subject must not have lesions requiring treatment in both the LAD and a diagonal branch.
2. Target lesion must be located in a native coronary artery with a visually estimated or quantitatively assessed %DS of ≥ 50% and < 100% with a thrombolysis in myocardial infarction (TIMI) flow of ≥ 1 and one of the following: stenosis ≥ 70%, an abnormal functional test (e.g., fractional flow reserve, stress test), unstable angina or post-infarct angina.
3. Target lesion must have a Dmax (by on-line QCA) or reference vessel diameter (RVD) (by visual estimation) ≥ 2.50 mm and ≤ 3.75 mm (on-line QCA assessment is recommended).
4. Target lesion must have a lesion length ≤ 24 mm based on either visual estimation or on-line QCA.

Angiographic Exclusion Criteria

All exclusion criteria apply to the target lesion(s) or target vessel(s). All exclusion criteria are based on visual estimation.

1. Target lesion is located in left main.
2. Aorto-ostial RCA target lesion (within 3 mm of the ostium).
3. Target lesion located within 3 mm of the origin of the LAD or LCX.
4. Lesion involving a bifurcation with a:

   1. Side branch ≥ 2 mm in diameter, or
   2. Side branch with diameter stenosis ≥ 50%, or
   3. Side branch requiring protection guide wire, or
   4. Side branch requiring pre-dilatation
5. Anatomy proximal to or within the lesion that may impair delivery of the Absorb BVS or XIENCE V, including:

   1. Extreme angulation (≥ 90°) proximal to or within the target lesion
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion
   3. Moderate or heavy calcification proximal to or within the target lesion
6. Target lesion or target vessel involves a myocardial bridge.
7. Target vessel contains thrombus as indicated in the angiographic images.
8. Target vessel has been previously treated with a stent at any time prior to the index procedure such that the Absorb BVS or XIENCE V would need to cross the stent to reach the target lesion.
9. Target vessel has been previously treated with a stent and the target lesion is within 5 mm proximal to a previously treated lesion.
10. Target lesion which prevents complete balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

    1. Residual %DS is < 40% (per visual estimation), ≤ 20% is strongly recommended.
    2. TIMI Grade-3 flow (per visual estimation).
    3. No angiographic complications (e.g. distal embolization, side branch closure).
    4. No dissections National Heart, Lung, and Blood Institute (NHLBI) grade D-F.
    5. No chest pain lasting > 5 minutes.
    6. No ST depression or elevation lasting > 5 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gao Runlin, MD, FACC, Principal Investigator — Fu Wai Hospital
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- [Derived] Stone GW, Kimura T, Gao R, Kereiakes DJ, Ellis SG, Onuma Y, Chevalier B, Simonton C, Dressler O, Crowley A, Ali ZA, Serruys PW. Time-Varying Outcomes With the Absorb Bioresorbable Vascular Scaffold During 5-Year Follow-up: A Systematic Meta-analysis and Individual Patient Data Pooled Study. JAMA Cardiol. 2019 Dec 1;4(12):1261-1269. doi: 10.1001/jamacardio.2019.4101. PMID 31561250
- [Derived] Ali ZA, Gao R, Kimura T, Onuma Y, Kereiakes DJ, Ellis SG, Chevalier B, Vu MT, Zhang Z, Simonton CA, Serruys PW, Stone GW. Three-Year Outcomes With the Absorb Bioresorbable Scaffold: Individual-Patient-Data Meta-Analysis From the ABSORB Randomized Trials. Circulation. 2018 Jan 30;137(5):464-479. doi: 10.1161/CIRCULATIONAHA.117.031843. Epub 2017 Oct 31. PMID 29089314
- [Derived] Stone GW, Gao R, Kimura T, Kereiakes DJ, Ellis SG, Onuma Y, Cheong WF, Jones-McMeans J, Su X, Zhang Z, Serruys PW. 1-year outcomes with the Absorb bioresorbable scaffold in patients with coronary artery disease: a patient-level, pooled meta-analysis. Lancet. 2016 Mar 26;387(10025):1277-89. doi: 10.1016/S0140-6736(15)01039-9. Epub 2016 Jan 27. PMID 26825231
- [Derived] Gao R, Yang Y, Han Y, Huo Y, Chen J, Yu B, Su X, Li L, Kuo HC, Ying SW, Cheong WF, Zhang Y, Su X, Xu B, Popma JJ, Stone GW; ABSORB China Investigators. Bioresorbable Vascular Scaffolds Versus Metallic Stents in Patients With Coronary Artery Disease: ABSORB China Trial. J Am Coll Cardiol. 2015 Dec 1;66(21):2298-2309. doi: 10.1016/j.jacc.2015.09.054. Epub 2015 Oct 12. PMID 26471805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of the ABSORB China RCT began on July 31, 2013 & completed on March 13, 2014 with the first subject randomized on 2 August 2013. A total of 480 subjects (Intent-to-treat (ITT) population) were randomized (Absorb BVS:241&XIENCE:239) at 24 clinical sites in mainland China. Last subject completed the 5 year follow-up on March 7, 2019.
Pre-assignment Details: Of the 480 ITT subjects, 21 were excluded from the PTE population due to pre-specified protocol/treatment deviations or due to subject withdrawal prior to any study device attempts during the index procedure. Thus, of the 459 subjects in the PTE population, 227 were randomized to the Absorb BVS arm and 232 were randomized to the XIENCE V arm
Period: Overall Study
Arm/Group | Absorb BVS System | XIENCE V EECSS
Started | 227 | 232
Completed | 221 | 223
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 4 | 9
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorb BVS System | XIENCE V EECSS | Total
Number analyzed (Participants) | 227 | 232 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.4) | 57.7 (9.6) | 57.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 61 | 127
  Male | 161 | 171 | 332
Region of Enrollment [Count of Participants; unit: Participants]
  China | 227 | 232 | 459

OUTCOME MEASURES:

1. Primary Outcome: In-segment Late Loss (LL) - Per Subject Analysis
Description: In-segment late loss is defined as the change in minimal lumen diameter (MLD) within the margins of the scaffold/stent and 5 mm proximal and 5 mm distal to the scaffold/stent from post-procedure to 1 year by angiography.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 196
Millimeter | 0.19 (0.38) | 0.13 (0.38)

2. Primary Outcome: In-segment Late Loss (LL) - Per Lesion Analysis
Description: as for outcome 1
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 196
Number analyzed (Target lesions) | 212 | 209
Millimeter | 0.19 (0.40) | 0.13 (0.37)

3. Secondary Outcome: Acute Device Success
Description: Successful delivery and deployment of the assigned scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final inscaffold/stent residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable). When bailout scaffold/stent is used, the success or failure of the bailout scaffold/stent delivery and deployment is not one of the criteria for device success.
  Acute success (device success and procedure success) was determined based on the device randomized while the Per-Treatment-Evaluable Population analysis must be based on the device actually received. Hence, device success and procedure success were provided for the ITT population only.
Time Frame: < or = 1 day
Population: Intent to treat set (ITT). Four subjects (1 in the Absorb BVS arm and 3 in the XIENCE V arm) were excluded from the data analysis for acute success.
  During the index procedure, 5 subjects withdrew consent following randomization and before any device attempts,3 in the Absorb BVS arm and 2 in the XIENCE V arm were excluded from all data analyses.
Measure: Number; unit: Percentage of target lesions
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 237 | 234
Number analyzed (Target lesions) | 250 | 249
Percentage of target lesions | 98.0 | 99.6

4. Secondary Outcome: Number of Participants With Acute Procedural Success
Description: Achievement of final in-scaffold/stent residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable) with successful delivery and deployment of at least one assigned scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay (maximum of 7 days). In dual target lesion setting, both lesions must meet clinical procedure success criteria to have a patient level procedure success.
  Acute success (device success and procedure success) was determined based on the device randomized while the Per-Treatment-Evaluable Population (PTE) analysis must be based on the device actually received. Hence, device success and procedure success were provided for the ITT population only.
Time Frame: At time of procedure up to 7 days in hospital
Population: ITT set. Four subjects (Absorb BVS (1) arm and XIENCE V arm (3)) were excluded from the data analysis for acute success. During the index procedure, 5 subjects withdrew consent following randomization and before any device attempts. Data from these 5 subjects (3 in the Absorb BVS arm and 2 in the XIENCE V arm) were excluded from all data analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 237 | 234
Participants | 230 | 230

5. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 0 | 0

6. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 0 to 37days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 0 | 0

7. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 0 | 3

8. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 0 | 4

9. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 0 | 4

10. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 1 | 5

11. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 2 | 5

12. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: as for outcome 5
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 4 | 7

13. Secondary Outcome: Number of Death (Cardiac, Vascular, Non-cardiovascular)
Description: Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 6 | 7

14. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: MI was categorized as Q-wave MI (QMI) and non-Q-wave MI (NQMI) and also MI attributable to target vessel (TV-MI) and MI not attributable to target vessel (NTV-MI). In addition, MIs were adjudicated based on three different MI definitions (per-protocol, modified ARC and WHO definitions) with the per-protocol analysis being the primary analysis for the study.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

15. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 0 to 37 days
Population: Per-Treatment-Evaluable Population. Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 3

16. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 4

17. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 4

18. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 3 | 4

19. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 5 | 5

20. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 6 | 5

21. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 7 | 6

22. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 14
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 7 | 6

23. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 0

24. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 0

25. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 4

26. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 1

27. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 7 | 7

28. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 9 | 8

29. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up..
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 11 | 8

30. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 12 | 9

31. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: * Ischemia-driven TLR (ID-TLR)
  * Not ischemia-driven TLR (NID-TLR)
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 12 | 9

32. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 0

33. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 0

34. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 1

35. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 1

36. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 9 | 12

37. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 11 | 13

38. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 14 | 13

39. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 16 | 16

40. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: * Ischemia-driven TVR (ID-TVR)
  * Not ischemia-driven TVR (NID-TVR)
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 16 | 16

41. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: All coronary revascularization includes percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG)
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 0

42. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 0 to 37days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 0

43. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 1

44. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 0 to 298 Days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 2

45. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 16 | 17

46. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 2 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 21 | 20

47. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 24 | 21

48. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 27 | 26

49. Secondary Outcome: Number of Participants With All Coronary Revascularization (PCI and CABG)
Description: as for outcome 41
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 28 | 26

50. Secondary Outcome: Number of Death/All MI
Description: All deaths includes Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Those MIs which are not Q-wave MI
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

51. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 3

52. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 6

53. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 6

54. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 3 | 6

55. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 6 | 8

56. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 8 | 8

57. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 11 | 10

58. Secondary Outcome: Number of Death/All MI
Description: as for outcome 50
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 13 | 10

59. Secondary Outcome: Number of Cardiac Death/All MI
Description: Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

60. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 3

61. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 4

62. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 4

63. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 3 | 4

64. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 6 | 5

65. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 7 | 5

66. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 9 | 6

67. Secondary Outcome: Number of Cardiac Death/All MI
Description: as for outcome 59
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 10 | 6

68. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

69. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 3

70. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 7

71. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 8

72. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 17 | 22

73. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 22 | 26

74. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up..
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 26 | 27

75. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 31 | 34

76. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 34 | 34

77. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: Target lesion failure (TLF) composite of Cardiac Death, Myocardial Infarction attributable to Target Vessel (TV-MI), or Ischemia-Driven Target Lesion Revascularization (ID-TLR))
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

78. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 2

79. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 4

80. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 5

81. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 7 | 9

82. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 9 | 10

83. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 12 | 10

84. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 15 | 12

85. Secondary Outcome: Number of Participants With Cardiac Death/TV-MI/ID-TLR [Target Lesion Failure (TLF)]
Description: as for outcome 77
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 16 | 12

86. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: ≤ 7 days post index procedure (In-hospital)
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

87. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 3

88. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 5

89. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 5

90. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 8 | 13

91. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 11 | 15

92. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 14 | 15

93. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up..
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 18 | 19

94. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TVR [Target Vessel Failure (TVF)]
Description: as for outcome 86
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 19 | 19

95. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and Ischemic driven target lesion revascularization (ID-TLR).
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 1 | 2

96. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 0 to 37 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 2 | 3

97. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 0 to 208 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 5

98. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 0 to 298 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants | 3 | 5

99. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 232
Participants | 7 | 9

100. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 2 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up..
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 10 | 11

101. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 3 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 230
Participants | 13 | 11

102. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 4 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 230
Participants | 16 | 13

103. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Event [MACE])
Description: as for outcome 95
Time Frame: 5 years
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants | 17 | 13

104. Secondary Outcome: Number of Participants With Acute Stent/Scaffold Thrombosis (Per Academic Research Consortium (ARC) Definition)
Description: Stent thrombosis was defined by Academic Research Consortium (ARC) criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy), probable (any unexplained death within the first 30 days or, regardless of the time after the index procedure, any Myocardial infarction (MI) related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause), and possible (any unexplained death from 30 days after intracoronary stenting until end of trial follow-up). Stent thrombosis was categorized as acute (0-24 hours post stent implantation), Subacute (>24 hours to 30 days post stent implantation), late (>30 days to 1 year post stent implantation).
Time Frame: < or = 1 day
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants
  Definite | 0 | 0
  Probable | 0 | 0

105. Secondary Outcome: Number of Participants With Subacute Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: >1 to 30 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 227 | 232
Participants
  Definite | 0 | 0
  Probable | 1 | 0

106. Secondary Outcome: Number of Participants With Late Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 31 to 365 days
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 226 | 228
Participants
  Definite | 0 | 0
  Probable | 0 | 0

107. Secondary Outcome: Number of Participants With Very Late 1 to 2 Year Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 366 to 730 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 225 | 225
Participants
  Definite | 1 | 0
  Probable | 0 | 0

108. Secondary Outcome: Number of Participants With Very Late 2 to 3 Year Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 731 to 1095 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 223 | 225
Participants
  Definite | 0 | 0
  Probable | 0 | 0

109. Secondary Outcome: Number of Participants With Very Late 1 to 3 Year Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 366-1095 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 224 | 225
Participants
  Definite | 1 | 0
  Probable | 0 | 0

110. Secondary Outcome: Number of Participants With Very Late 3 to 4 Year Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 1096-1460 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 221 | 223
Participants
  Definite | 0 | 0
  Probable | 1 | 1

111. Secondary Outcome: Number of Participants With Very Late 4 to 5 Year Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 1461-1825 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 216 | 215
Participants
  Definite | 0 | 0
  Probable | 0 | 0

112. Secondary Outcome: Number of Participants With Very Late 3 to 5 Year Stent/Scaffold Thrombosis (Per ARC Definition)
Description: as for outcome 104
Time Frame: 1096-1825 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 217 | 216
Participants
  Definite | 0 | 0
  Probable | 1 | 1

113. Secondary Outcome: Over All Number of Participants With Cumulative 5 Year Stent /Scaffold Thrombosis
Description: as for outcome 104
Time Frame: 0-1825 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 218 | 216
Participants
  Definite | 1 | 0
  Probable | 2 | 1

114. Secondary Outcome: In-Device Minimum Lumen Diameter (MLD)
Description: Minimum lumen diameter is defined as the shortest diameter through the center point of the lumen. Data are collected from two projections.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 197
Number analyzed (Target lesions) | 212 | 210
Millimeter | 2.24 (0.48) | 2.50 (0.46)

115. Secondary Outcome: In-Segment Minimum Lumen Diameter (MLD)
Description: Minimum lumen diameter is defined as the shortest diameter through the center point of the lumen. Data are collected from two projections.
  INSEGMENT: Within the margins of the scaffold/stent and 5 mm proximal and 5 mm distal to the scaffold/stent.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 197
Number analyzed (Target lesions) | 212 | 210
Millimeter | 2.11 (0.47) | 2.17 (0.49)

116. Secondary Outcome: Proximal Minimum Lumen Diameter (MLD)
Description: as for outcome 114
Time Frame: 1 year
Population: Per-Treatment-Evaluable Population (PTE) Population. Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 198 | 192
Number analyzed (Target lesions) | 208 | 205
Millimeter | 2.64 (0.48) | 2.68 (0.56)

117. Secondary Outcome: Distal Minimum Lumen Diameter (MLD)
Description: as for outcome 114
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 199 | 196
Number analyzed (Target lesions) | 210 | 209
Millimeter | 2.39 (0.45) | 2.37 (0.50)

118. Secondary Outcome: In-Segment Percent Diameter Stenosis (%DS)
Description: The Percent Diameter Stenosis value calculated as 100 * (1 MLD/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA). Reference vessel diameter based on QCA is derived from either the user defined method using average diameter of proximal and distal healthy segments or the interpolated method.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 197
Number analyzed (Target lesions) | 212 | 210
Percent Diameter stenosis | 24.02 (13.23) | 22.96 (13.18)

119. Secondary Outcome: In-Device Percent Diameter Stenosis (%DS)
Description: as for outcome 118
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 197
Number analyzed (Target lesions) | 212 | 210
Percent Diameter stenosis | 19.16 (14.36) | 11.15 (11.38)

120. Secondary Outcome: Proximal Percent Diameter Stenosis (%DS)
Description: as for outcome 118
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 198 | 192
Number analyzed (Target lesions) | 208 | 205
Percent Diameter stenosis | 11.09 (10.13) | 12.12 (11.63)

121. Secondary Outcome: Percentage of Participants With Proximal Angiographic Binary Restenosis (ABR)
Description: Angiographic Binary Restenosis (ABR): Renarrowing of the artery defined as %DS ≥ 50%.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 198 | 192
Number analyzed (Target lesions) | 208 | 205
Percentage of participants | 1.0 | 1.5

122. Secondary Outcome: Distal Percent Diameter Stenosis (%DS)
Description: as for outcome 118
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 199 | 196
Number analyzed (Target lesions) | 210 | 209
Percent Diameter stenosis | 8.53 (8.15) | 8.14 (11.86)

123. Secondary Outcome: Percentage of Participants With In-Segment Angiographic Binary Restenosis (ABR)
Description: Angiographic Binary Restenosis (ABR): Renarrowing of the artery defined as %DS ≥ 50%. InSegment is defined as within the margins of the scaffold/stent and 5 mm proximal and 5 mm distal to the scaffold/stent.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 197
Number analyzed (Target lesions) | 212 | 210
percentage of participants | 4.2 | 2.9

124. Secondary Outcome: Percentage of Participants With In-Device Angiographic Binary Restenosis (ABR)
Description: Angiographic Binary Restenosis (ABR): Renarrowing of the artery defined as %DS ≥ 50%.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 197
Number analyzed (Target lesions) | 212 | 210
Percentage of participants | 3.3 | 1.0

125. Secondary Outcome: In-Segment Late Loss (LL)
Description: In-segment Late Loss is calculated as (in-segment MLD post-procedure) - (in-segment MLD at followup).
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 196
Number analyzed (Target lesions) | 212 | 209
Millimeter | 0.19 (0.40) | 0.13 (0.37)

126. Secondary Outcome: Percentage of Participants With Distal Angiographic Binary Restenosis (ABR)
Description: Angiographic Binary Restenosis (ABR): Renarrowing of the artery defined as %DS ≥ 50%.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 199 | 196
Number analyzed (Target lesions) | 210 | 209
Percentage of participants | 0.0 | 1.0

127. Secondary Outcome: In-Device Late Loss (LL)
Description: In-device late loss is calculated as (in-device MLD post-procedure) - (in-device MLD at followup).
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 200 | 196
Number analyzed (Target lesions) | 212 | 209
Millimeter | 0.24 (0.39) | 0.10 (0.32)

128. Secondary Outcome: Proximal Late Loss (LL)
Description: Proximal Late Loss: Proximal MLD post procedure - Proximal MLD at followup.
  Proximal is defined as within 5 mm of healthy tissue proximal to the device placement.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 196 | 185
Number analyzed (Target lesions) | 205 | 198
Millimeter | 0.19 (0.39) | 0.13 (0.42)

129. Secondary Outcome: Distal Late Loss (LL)
Description: Distal Late Loss calculated as Distal MLD post procedure - Distal MLD at followup.
  Distal is defined as within 5 mm of healthy tissue distal to the device placement.
Time Frame: 1 year
Population: Per-Treatment Evaluable Population set (PTE). Analysis population exclude subjects who are truly lost-to-follow-up.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS System | XIENCE V EECSS
Number analyzed (Participants) | 199 | 194
Number analyzed (Target lesions) | 210 | 207
Millimeter | 0.08 (0.31) | 0.03 (0.33)

ADVERSE EVENTS:
Time Frame: 5 years
Description: PTE population.
Arm/Group | Absorb BVS System | XIENCE V EECSS
All-Cause Mortality (participants affected / at risk) | 6/227 | 7/232
Serious Adverse Events (participants affected / at risk) | 94/227 | 81/232
Other Adverse Events (participants affected / at risk) | 151/227 | 135/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS System (N=227) | XIENCE V EECSS (N=232)
Atrial fibrillation (Cardiac disorders) | 2 | 2
Coronary artery dissection (Cardiac disorders) | 4 | 5
Coronary artery stenosis (Cardiac disorders) | 10 | 8
Myocardial infarction (Cardiac disorders) | 4 | 2
Palpitations (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Hematochezia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Application site hematoma (General disorders) | 1 | 0
Chest discomfort (General disorders) | 8 | 5
Chest pain (General disorders) | 2 | 1
Drug resistance (General disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 9 | 11
Electric injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 12 | 5
Angina unstable (Cardiac disorders) | 15 | 10
Cardiac failure (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 11 | 4
Extrasystoles (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (Gastrointestinal disorders) | 0 | 1
Mass (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 4
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram coronary (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Physical examination (Investigations) | 0 | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 2
Lacunar infarction (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Intestinal Polyp (Gastrointestinal disorders) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Neuromyelitis Optica (Nervous system disorders) | 1 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS System (N=227) | XIENCE V EECSS (N=232)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 28 | 16
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Coronary artery dissection (Cardiac disorders) | 4 | 5
Coronary artery stenosis (Cardiac disorders) | 10 | 8
Coronary artery disease (Cardiac disorders) | 12 | 4
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 4 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 4
Extrasystoles (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 16 | 12
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Hematochezia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 3
Application site haematoma (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Chest discomfort (General disorders) | 25 | 14
Non-cardiac chest pain (General disorders) | 8 | 11
Chest pain (General disorders) | 2 | 2
Irritability (General disorders) | 1 | 0
Drug resistance (General disorders) | 1 | 0
Mass (General disorders) | 0 | 1
Sensation of foreign body (General disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 4 | 2
Lung infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 9 | 11
Electric injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Cardiac enzymes increased (Investigations) | 10 | 9
Blood creatine phosphokinase MB increased (Investigations) | 7 | 4
Blood creatine phosphokinase increased (Investigations) | 5 | 4
Blood creatinine increased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 25 | 32
Troponin T increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Brain oedema (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 3
Hemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Xerophthalmia (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram coronary (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Physical examination (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Intestinal Polyp (Gastrointestinal disorders) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Neuromyelitis Optica (Nervous system disorders) | 1 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less